CLINICAL TRIAL: NCT03542682
Title: The Effect of Insulin Bolus Speed of Rapid-Acting Insulin Analog Absorption and Action in Individuals With Type 1 Diabetes
Brief Title: The Effect of Bolus Speed of Rapid-Acting Insulin Analog Absorption and Action in Individuals With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000022726
Record Dates: First submitted 2018-04-30; First posted 2018-05-31 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Type1diabetes

STUDY DESIGN:
Intervention Model Description: This study will be a cross-over, randomized order, single blinded clinical study in subjects with Type 1 Diabetes.
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Individuals given Standard Bolus first, then quick bolus (Active Comparator): Individuals with Type 1 Diabetes (T1D) will receive both Standard and Quick Bolus in a randomized cross-over design.
  Interventions: Device: Quick Bolus; Device: Standard Bolus
- Individuals given Quick bolus first, then standard bolus (Active Comparator): Individuals with Type 1 Diabetes (T1D) will receive both Standard and Quick Bolus in a randomized cross-over design.
  Interventions: Device: Quick Bolus; Device: Standard Bolus

INTERVENTIONS:
Device: Quick Bolus — Individuals with Type 1 Diabetes (T1D) given 0.2 units/kg of rapid acting insulin (RAI) via "quick bolus" of 15 units per minute during a euglycemic clamp.
Device: Standard Bolus — Individuals with Type 1 Diabetes (T1D) given 0.2 units/kg of rapid acting insulin (RAI) via "standard bolus" of 1.5 units per minute during a euglycemic clamp.

SUMMARY:
Rapid Action Insulin (RAI) absorption and action measured by time to reach maximum insulin concentration and glucose infusion rate.

DETAILED DESCRIPTION:
The investigators hypothesize that RAI absorption and action measured by time to reach maximum insulin concentration and glucose infusion rate during the clamp study will be significantly faster when insulin bolus is delivered using the "Quick Bolus" feature as compared to the "Standard Bolus".

Outcomes were updated at time of results entry.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 30 (inclusive)
2. Clinical diagnosis of T1D of at least one year's duration
3. On Continuous Subcutaneous Insulin Infusion (CSII) therapy for at least three months
4. HbA1c <10%
5. Minimum weight requirement of at least 37.9 kg
6. Ability to comprehend written and spoken English
7. Total daily requirement of insulin between 0.6 and1.2 U/kg/day
8. Not have any other medical condition or disease known to affect insulin action and glucose control aside from T1D or treated hypothyroidism

Exclusion Criteria:

1. Medication besides insulin known to alter blood glucose or insulin action
2. Female subjects of reproductive potential that are pregnant or breast feeding, or not consistently using a barrier method or abstinence as contraception.
3. Inability to comprehend written and spoken English
4. Any other condition, which in the judgment of the investigators, would interfere with the subject's ability to provide informed consent or the investigator's ability to perform the study
5. Hematocrit less than 35% or a serum potassium less than 3.4 mmol/L

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eda Cengiz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants consented to participate but 2 were lost to follow up prior to randomization
Period: Overall Study
Arm/Group | Individuals Given Standard Bolus First, Then Quick Bolus | Individuals Given Quick Bolus First, Then Standard Bolus
Started (Participants randomized) | 5 | 4
Completed First Stage | 5 | 4
Completed Second Stage | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 1
Not completed — COVID-19 Protocol | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographics were collected from the 8 who completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Individuals Given Standard Bolus First, Then Quick Bolus | Individuals Given Quick Bolus First, Then Standard Bolus | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (3.3) | 20.7 (3.1) | 22 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Baseline mean percent Hemoglobin A1c [Mean (Standard Deviation); unit: percent Hemoglobin A1c] | 7.6 (1.3) | 7.9 (1.1) | 7.7 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximum Glucose Infusion Rate
Description: time to maximum glucose infusion rate (GIR) in minutes
Time Frame: 300 minutes
Population: Complete case analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Quick Bolus | Standard Bolus
Number analyzed (Participants) | 8 | 8
minutes | 116.54 [74.74 to 158.34] | 172.21 [130.41 to 214.01]
Statistical Analysis 1: Comparison: Quick Bolus vs Standard Bolus; Test type: Superiority; Mixed Models Analysis; The model adjusted for order of the clamps and accounting for within subject correlation; Mean Difference (Final Values) = -55.67, 95% CI 2-sided [-124.63 to 13.30]

2. Secondary Outcome: Earlier Clearance of Exogenous Insulin.
Description: Time to reach baseline insulin concentrations is used to determine the completion of insulin as part bolus of bioavailability.
Time Frame: up to 5 hours
Population: Outcome was not part of the study protocol and therefore was not collected.
Arm/Group | Standard Bolus | Quick Bolus
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Maximum Glucose Infusion Rate
Description: maximum glucose infusion rate (GIRmax)
Time Frame: 300 minutes
Population: Complete case analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/kg/min
Arm/Group | Quick Bolus | Standard Bolus
Number analyzed (Participants) | 8 | 8
mg/kg/min | 8.42 [4.91 to 11.92] | 7.45 [3.95 to 10.96]
Statistical Analysis 1: Comparison: Quick Bolus vs Standard Bolus; Test type: Superiority; Mixed Models Analysis; The model adjusted for order of the clamps and accounting for within subject correlation; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-1.10 to 3.02]

4. Secondary Outcome: Area Under the Curve for the Glucose Infusion Rate
Description: area under the curve for the glucose infusion rate
Time Frame: 300 minutes
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Quick Bolus | Standard Bolus
Number analyzed (Participants) | 8 | 8
mg/kg | 1204.29 [716.72 to 1691.86] | 1072.44 [584.86 to 1560.01]
Statistical Analysis 1: Comparison: Quick Bolus vs Standard Bolus; Test type: Superiority; Mixed Models Analysis; The model adjusted for order of the clamps and accounting for within subject correlation; Mean Difference (Final Values) = 131.85, 95% CI 2-sided [-246.70 to 510.41]

ADVERSE EVENTS:
Time Frame: Up to 5 hours post intervention for each intervention
Groups:
- Individuals Given Standard Bolus: Individuals with Type 1 Diabetes (T1D) will receive both Standard and Quick Bolus in a randomized cross-over design.
  Standard Bolus: Individuals with Type 1 Diabetes (T1D) given 0.2 units/kg of rapid acting insulin (RAI) via "standard bolus" of 1.5 units per minute during a euglycemic clamp.
- Individuals Given Quick Bolus: Individuals with Type 1 Diabetes (T1D) will receive both Standard and Quick Bolus in a randomized cross-over design.
  Quick Bolus: Individuals with Type 1 Diabetes (T1D) given 0.2 units/kg of rapid acting insulin (RAI) via "quick bolus" of 15 units per minute during a euglycemic clamp.
Arm/Group | Individuals Given Standard Bolus | Individuals Given Quick Bolus
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individuals Given Standard Bolus (N=8) | Individuals Given Quick Bolus (N=9)
Common Cold (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT03542682/Prot_SAP_000.pdf